CLINICAL TRIAL: NCT00015886
Title: Docetaxel (Taxotere) and 5-Fluorouracil As Second- Or Third-Line Chemotherapy In Women With Metastatic Breast Cancer
Brief Title: Combination Chemotherapy in Treating Women With Breast Cancer That is Metastatic or Cannot be Treated With Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068567; CCCWFU-74896; NCI-3137
Record Dates: First submitted 2001-05-06; First posted 2003-10-15 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: docetaxel — 75 milligrams per meter squared intraveneously
Drug: fluorouracil — 350 milligrams intraveneously

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating women who have breast cancer that is metastatic or cannot be treated with surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in women with locally unresectable or metastatic breast cancer treated with docetaxel, leucovorin calcium, and fluorouracil as second or third-line chemotherapy.
* Evaluate the toxic effects of this regimen in these patients.
* Determine the time to progression in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour on day 1 and leucovorin calcium IV over 1 hour followed by fluorouracil IV over 5 minutes on days 1-3. Treatment repeats every 4 weeks for 2-8 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 21-45 patients will be accrued for this study within 44 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic or unresectable local disease
* Measurable or evaluable disease
* No ascites or pleural effusion as only metastatic site
* No brain or leptomeningeal metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Granulocyte count greater than 1,500/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Bilirubin normal
* SGOT/SGPT less than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 2.5 times ULN

Renal:

* Creatinine no greater than 2 times ULN

Cardiovascular:

* Adequate cardiac function
* No history of significant atherosclerotic coronary disease (e.g., uncontrolled angina)
* No history of significant cardiac arrhythmia

Other:

* No serious medical or psychiatric illness that would preclude study
* No active uncontrolled bacterial, viral, or fungal infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior high-dose chemotherapy and autologous transplantation

Chemotherapy:

* At least 3 weeks since prior chemotherapy and recovered
* No more than 2 prior chemotherapy regimens for metastatic breast cancer (in addition to adjuvant therapy)
* No prior docetaxel
* No prior high-dose chemotherapy and autologous transplantation
* Prior paclitaxel allowed

Endocrine therapy:

* No concurrent hormonal therapy, except as contraception

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered
* Concurrent radiotherapy for relief of localized pain or obstruction allowed

Surgery:

* At least 2 weeks since prior major surgery and recovered

Other:

* No other concurrent cytotoxic agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1997-01; Primary Completion 2002-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
To determine the response rate to this combination after two to four courses of Docetaxel (Taxotere) And 5-Fluorouracil | 28 weeks

SECONDARY OUTCOMES:
To evaluate toxicities of Docetaxel (Taxotere) And 5-Fluorouracil | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Kimmick, MD, MS, Study Chair — Wake Forest University Health Sciences
Locations (6):
- United States (6):
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Palmetto Hematology/Oncology Associates, Spartanburg, South Carolina
  - Massey Cancer Center, Richmond, Virginia